CLINICAL TRIAL: NCT04449809
Title: Pilot Study of the Feasibility of an Exercise Regimen Designed to Improve Functional Mobility, Body Composition, and Strength After Breast Conservation Therapy for Women With Early Stage Breast Cancer
Brief Title: Exercise Regimen Designed to Improve Functional Mobility, Body Composition, and Strength After Breast Conservation Therapy for Women With Early Stage Breast Cancer
Acronym: EXERT-BC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll due to COVID-19
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104863
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Exercise program
  Interventions: Behavioral: Exercise program

INTERVENTIONS:
Behavioral: Exercise program — 3x per week group monitored group exercise sessions

SUMMARY:
The purpose of this research study is to find out if a monitored group exercise program can increase strength, muscle mass and ability to move in women after treatment for early stage breast cancer.

DETAILED DESCRIPTION:
This trial will assess the safety and feasibility of a monitored group exercise regimen utilizing high-load resistance training and functional exercises with compound movements in a group of women treated for early stage breast cancer with the goal of improving functional mobility, body composition, and strength after breast conservation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-70 years
2. Women with a biopsy proven diagnosis of ductal carcinoma in situ or invasive carcinoma of the breast
3. Women must have undergone breast conservation therapy with no neoadjuvant or adjuvant chemotherapy (adjuvant endocrine therapy is permitted)
4. BMI > 25 kg/m2 or body fat% greater or equal to 31%
5. Participants must have abstained from smoking for at least 12 months
6. Women of child-bearing potential must verbally confirm lack of pregnancy prior to enrollment and have undergone a pregnancy test prior to initial of radiation therapy (standard protocol for radiation therapy). They should also consent to use adequate contraception during the course of the study.
7. Women must be determined capable of engaging in resistance training as documented in treating radiation oncologist notes.
8. Participants must have a schedule amenable to three prescheduled workout sessions per week, scheduled during the day.
9. Women must complete a Functional Mobility Screen (FMS) and determined safe to engage in the workout regimen by the study personnel.

Exclusion Criteria:

1. Any treatment with chemotherapy for recent breast cancer treatment
2. Mastectomy and/or lymph node dissection
3. Uncontrolled hypertension or diabetes, defined as systolic blood pressure over 149, diastolic blood pressure over 99, and hemoglobin A1c greater than 8.9.
4. Diabetic condition requiring the usage of insulin
5. Severe arthritic, joint, cardiovascular, or musculoskeletal condition
6. Inability to perform body weight squat exercise without pain assessed by treating radiation oncologist
7. History of myocardial infarction or coronary artery disease

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Adherence, defined as the proportion of participants completing at least 75% of the planned exercise sessions | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, MD CSCS, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No